CLINICAL TRIAL: NCT01571934
Title: Inhibitor Development in Patients With Hemophilia A Undergoing Surgery
Acronym: PASs
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christine Kempton, MD, MSc, Christine Kempton, MD, MSc, Emory University
Other Study IDs: IRB00046800; 5K23HL105785 (NIH); PASs (Other: Other)
Record Dates: First submitted 2012-04-04; First posted 2012-04-05 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood drawn during study includes 15 ml within 7 days prior to surgery and 15 ml drawn on post-operative days 1, 14 and 90.
  Samples for DNA storage will be generated from blood draw study samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild or moderate hemophilia A: Subjects with mild or moderate hemophilia A (fVIII activity 1-40%) who are scheduled to undergo surgery for which at least 5 consecutive days of fVIII replacement therapy is required.

SUMMARY:
Hemophilia A is a genetic deficiency of factor VIII that causes blood to clot too slowly. The disease is classified based on how much factor VIII is in the blood. People with mild or moderate hemophilia A have low, but detectable, blood levels of factor VIII and bleed with trauma or surgery. At the time of surgery, they need to receive factor VIII replacement by infusion into the vein so that blood can clot normally and abnormal bleeding can be avoided. A complication of hemophilia A is the development of an antibody that binds factor VIII and makes the factor VIII infused for treatment not work properly. This antibody is called an inhibitor. In mild and moderate hemophilia A, inhibitors are not common, but have been reported to occur after intensive factor VIII infusions, as may occur at the time of surgery. This study is designed to observe people with mild and moderate hemophilia A who are having surgery. Information on the surgery, treatments given, bleeding, and infection will be gathered. Also, blood will be drawn to determine how the immune system is reacting to the factor VIII. No specific treatments will be given as part of this study. We will use the information to determine what influences inhibitor development. A better understanding of inhibitor development will help medical providers do things to avoid inhibitor development in this population or researchers to design new treatments.

DETAILED DESCRIPTION:
The development of neutralizing anti-factor VIII (fVIII) antibodies, fVIII inhibitor, is the most significant complication affecting patients with hemophilia A (HA). Once an inhibitor develops, treatment is less effective and costly. Although inhibitors occur most commonly in those with severe HA, 25% of new inhibitors occur in those with non-severe HA. In patients with non-severe HA, the development of a fVIII inhibitor can change the course of disease from one that is easily managed to one with the potential for spontaneous life-threatening difficult to treat bleeding. Although significant advances have been made in understanding risk factors for fVIII inhibitor development in patients with severe HA, studies that seek to understand the risk for fVIII inhibitor development in those with non-severe disease have been limited to retrospective analyses. In these retrospective analyses, intensive fVIII treatment and surgery have been identified as risk factors for fVIII inhibitor development in non-severe HA. Additionally, receiving fVIII by continuous infusion has been associated with fVIII inhibitor development in non-severe HA in some but not all studies and may be due in part to a more robust proinflammatory response during continuous infusion. Accordingly, the next logical step to evaluate the risk of inhibitor development associated with continuous fVIII infusion is a prospective observational cohort study. Additionally, knowledge of the immune response to fVIII in the surgical setting is essential for identification of patients at high risk for inhibitor development and development of strategies to prevent inhibitor development and is best evaluated in the setting of an prospective cohort study.

This multicenter prospective observational cohort study will enroll a total of 140 subjects at 10 centers who have mild or moderate hemophilia a (fVIII activity 1-40%) who are scheduled to undergo surgery for which at least 5 consecutive days of fVIII replacement therapy is required. The study will gather clinical data and collect blood specimens on 4 occasions over a 3 month period. Outcomes include: inhibitor development, total fVIII usage, bleeding, and markers of T cell activation.

ELIGIBILITY:
Inclusion Criteria:

* Males with mild/moderate hemophilia A (fVIII activity 1-40%)
* Planned surgical intervention which is anticipated to require 5 consecutive days of fVIII replacement therapy (These can be outpatient or inpatient treatment days.)
* Weight >22.5 kg (To assure that volumes of blood to be drawn for study purposes are safe.)

Exclusion Criteria:

* Past history of an inhibitor (inhibitor titer >0.4 BU/ml)
* HIV infection with CD4 count <400/ul
* Currently receiving immunosuppressive medication(s)
* Unable to tolerate quantity of blood to be drawn
* Current or past diagnosis autoimmune disorder
* Current or past diagnosis of immune deficiency disorder other than HIV

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In addition to Emory University, subjects will be recruited at one of 8 following sites: University of Pittsburgh, University of North Carolina, Oregon Health and Science University, University of Colorado, University of Texas Health Science Center at Houston, University of Minnesota, and Indiana Hemophilia Treatment Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Inhibitor development (inhibitor titer > 0.4 BU/ml) | postopereratvie date 90
  Primary Study Endpoint: Inhibitor development (inhibitor titer > 0.4 BU/ml) by post-operative (POD) day 90. Three months or 90 days was selected as the primary end point based on data collected in the case-control study where 17/18 cases had developed their inhibitor within 12 weeks of their intensive fVIII treatment and only 1 case developed the inhibitor >16 weeks after the intensive fVIII treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kempton, MD, MSc, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - University of Colorado, Hemophilia and Thrombosis Center, Aurora, Colorado
  - Emory University Comprehensive Hemophilia Treatment Center, Atlanta, Georgia
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh and Hemophilia Center of Pennsylvania, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided